CLINICAL TRIAL: NCT00285870
Title: Quantification of Upper Extremity Hypertonia
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Terence Sanger, Associate Professor, University of Southern California
Other Study IDs: UPPER EXTREMITY HYPERTONIA
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Dystonia; Muscle Hypertonia
MeSH Terms: conditions — Dystonia; Muscle Hypertonia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Dr. Sanger and the research team want to learn about upper extremity hypertonia (stiffness) in children and young adults with cerebral palsy. Specifically, they want to learn about ways to measure the stiffness in the joints of hypertonic arms. The information the research team will collect includes any physical exams or computer generated data about your arm movements.

ELIGIBILITY:
Inclusion Criteria:Dystonia in at least one arm Age 4 to no upper limit

Exclusion Criteria:increased risk of participation botulinum toxin within 6 months

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children with cerebral palsy and/or dystonia.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Observation | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Terence D. Sanger, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States